CLINICAL TRIAL: NCT06366347
Title: A Phase 2 Trial of Maintenance Abemaciclib/Letrozole After Systemic Therapy in Patients With Advanced or Recurrent Estrogen Receptor Positive, Mismatch Repair Proficient, TP53 Wildtype Endometrial Cancer
Brief Title: ALPINE: Maintenance Letrozole/Abemaciclib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Panagiotis Konstantinopoulos, MD, PhD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-695
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer; Recurrent Endometrial Cancer; TP53
Keywords: TP53 wild-type endometrial cancer; Endometrial Cancer; Recurrent endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — abemaciclib; Letrozole; pembrolizumab; Antibodies, Monoclonal; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1: Abemaciclib + Letrozole (Experimental): Participants will be stratified by Primary Stage IVb (4b) vs. Primary Measurable Stage III (3)/IVa (4a) vs. Recurrent Endometrial Cancer and will complete study procedures as follows:
  * Baseline visit with X-ray, CT, MRI, or PET scan.
  * Cycles 1 through 3:
    --Days 1 through 21 of 21 day cycle: Predetermined dose of Abemaciclib 2x per day. Predetermined dose of Letrozole 1x per day.
  * Cycle 4 and every 2 cycles thereafter:
    --Days 1 through 21 of 21 day cycle: Predetermined dose of Abemaciclib 2x per day. Predetermined dose of Letrozole 1x per day.
  * X-ray, CT, MRI, or PET scan every 9 weeks for first 9 months, then every 12 months.
  * End of Treatment visit with assessments and X-ray, CT, MRI, or PET scan.
  * Follow up for up to 3 years.
  Interventions: Drug: Abemaciclib; Drug: Letrozole; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Abemaciclib — CDK inhibitor, tablet taken orally per protocol.
  Other Names: Verzenio; LY2835219; C27H32F2N8
Drug: Letrozole — Aromatase inhibitor, tablet taken orally per protocol.
  Other Names: Femara; C17H11N5
Drug: Pembrolizumab — Humanized immunoglobulin G4 monoclonal antibody, 4mL (milliliter) single-dose vial, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Keytruda; MK-3475; Humanized X PD-1-mAB (monoclonal antibody) (H409A11) IgG4 (immunoglobulin G4); C6504H10004N1716O2036S46

SUMMARY:
The purpose of this research study is to see if the study drugs abemaciclib and letrozole are effective and safe for participants with estrogen-receptor positive (ER+), mismatch repair proficient, tumor protein p53 (TP53) wild-type endometrial cancer.

The names of the study drugs involved in this study are:

* Abemaciclib (a type of cyclin-dependent kinase (CDK) inhibitor)
* Letrozole (a type of aromatase inhibitor)

DETAILED DESCRIPTION:
This is a phase 2, single arm trial of maintenance letrozole/abemaciclib after carboplatin/paclitaxel chemotherapy with or without anti-PD-(L)1 blockade in patients with advanced or recurrent estrogen receptor (ER) positive (ER+), mismatch repair proficient (MMRP), tumor protein p53 (TP53) wild-type endometrial cancer.

The U.S. Food and Drug Administration (FDA) has not approved abemaciclib or letrozole for endometrial cancer but they have been approved for other uses.

The research study procedures include screening for eligibility, study treatment visits, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, blood tests, and electrocardiograms (EKGs).

Participants will be administered study drugs for up to 2 years and will be followed for 3 years after completing study treatment.

It is expected that about 32 people will take part in this research study.

Eli Lilly is supporting this research study by providing funding and the study drug abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed either i) endometrioid endometrial cancer or ii) endometrial carcinosarcoma with endometrioid epithelial component.
* Participants must have ER-positive disease, defined as ≥ 1 percent of tumor cell nuclei being immunoreactive by immunohistochemistry (IHC). If multiple analyses have been performed, judgment should be based on the most recent biopsy or pathology specimen analyzed in a CLIA (Clinical Laboratory Improvement Amendments)-certified laboratory.
* Tumor must be TP53 wild-type as determined by immunohistochemistry (IHC) or via CLIA-certified targeted Next-Generation Sequencing (NGS); IHC assessment of p53 status is included in the NCCN guidelines of uterine neoplasms for the molecular analysis of endometrial carcinoma.
* Participants must have mismatch repair proficient (MMRP) endometrial cancer as determined by immunohistochemistry (IHC) or polymerase chain reaction (PCR) or any CLIA-certified next generation sequencing assay.
* No known tumor mutational burden ≥ 10 mutations/megabase (Mb).
* No known RB1 mutations or two-copy RB1 deletion.
* Participants must have just completed a minimum of 4 cycles and a maximum of 10 cycles of a combination of carboplatin and taxane or a combination of taxane and anti-PD-(L)1 inhibitor therapy (e.g., pembrolizumab, or dostarlimab, or durvalumab).
* Participants must have had measurable stage III, measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial cancer.
* Participants are permitted to have received:

  * a. Prior adjuvant chemotherapy (e.g., paclitaxel/carboplatin alone or as a component of concurrent chemotherapy and radiation therapy [with or without cisplatin])
  * b. Prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/paraaortic radiation therapy, intravaginal brachytherapy, and/or palliative radiation therapy. All radiation therapy must have been completed at least 4 weeks prior to registration.
  * c. Prior hormonal therapy for treatment of endometrial cancer.
* Must be able to initiate study drug between 3 to 8 weeks (or 21 to 56 days) after completion of their final dose of chemotherapy and anti-PD-(L)1 blockade (if they were receiving anti-PD-(L)1 blockade).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (see Appendix A)
* Age ≥ 18 years
* Participants must have normal organ and bone marrow function within 2 weeks before starting protocol therapy as defined below:

  * System Laboratory Value
  * Hematologic

    * ANC ≥1.5 × 109 /L
    * Platelets ≥100 × 109 /L
    * Hemoglobin ≥8 g/dL Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Hepatic

    * Total bilirubin ≤1.5 × ULN Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
    * ALT and AST ≤3 × ULN
    * Creatinine ≤ 1.5 × institutional ULN, OR
    * Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 x institutional ULN.
    * Abbreviations: ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; ULN = upper limit of normal.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.
* Participants must be willing to release archival tissue if available. Please see section 9.1.2 and the laboratory manual for tissue requirements.

Exclusion Criteria:

* Participants who have received previous treatment with CDK4/6 inhibitors, including but not limited to previous abemaciclib therapy.
* Any gastrointestinal dysfunctions that could interfere with the absorption of study drugs (e.g., bowel obstruction, inability to swallow tablets, malabsorption syndrome, unresolved nausea, vomiting, diarrhea CTCAE v 5.0 > grade 1).
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to starting study treatment.
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* Major injuries or surgery within 14 days prior to start of study treatment and/or planned major surgery during the on-treatment study period. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and starting study treatment.
* Other malignant disease with disease-free ≤ 3 years except: curatively treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, or ductal carcinoma in situ (DCIS) of the breast or any other cancer deemed by the investigator to be at low risk for recurrence of that malignancy.
* Active brain metastases (e.g., stable for < 8 weeks, no adequate previous treatment with radiotherapy and/or surgery, symptomatic, requiring treatment with anti-convulsant therapy. Corticoid therapy is allowed if administered as stable dose for at least 1 month before starting study treatment).
* Females who are pregnant or lactating. The effects of the study agents on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of study agent. Contraceptive methods may include an intrauterine device (IUD) or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. A negative serum pregnancy test is required for study entry from women of childbearing potential.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease/pneumonitis, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Participants who at the time of study enrollment are known to require concomitant therapy with strong CYP3A4 inducers, or strong inhibitors of CYP3A4. Due to potential drug interactions, concomitant use of these medications is not permitted for the duration of treatment on trial. Participants are eligible for study entry if an appropriate substitution is made prior to the first dose of study medication.
* Participants with personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Individuals with a history of a different malignancy are ineligible with the following exceptions: individuals who have been treated and are disease-free for a minimum of 3 years prior to study enrollment, or individuals who are deemed by the treating investigator to be at low risk for disease recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date the participant was registered to the date of documented progressive disease (PD) by RECIST version 1.1 or death (regardless of cause) in the absence of progression, regardless of whether the participant withdraws from study drug or receives another anti-cancer therapy prior to progression. Participants alive without disease progression are censored at date of last disease evaluation. A participant who dies without progression, and the death is >12 weeks after the last evaluable tumor assessment, is censored for PFS at the date of last disease evaluation. A participant who has no baseline or no post treatment tumor assessment is censored at 0 days for PFS, unless she dies < 12 weeks from randomization, in which case the PFS event date is the death date. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum, taking as reference the smallest sum on study with at least 5 mm absolute increase.

SECONDARY OUTCOMES:
Grade 3-5 Adverse Events (AE) Rate | Up to 2 years and 1 month
  Grade 3-5 AE rate is defined as the proportion of patients who experience a grade 3-5 adverse event based on the Common Toxicity Criteria for Adverse Events version 5.0 as reported on case report form.
Median Overall Survival (OS) | Up to 5 years
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive based on Kaplan-Meier methodology.
Objective Response Rate (ORR) | Up to 2 years
  The percentage of participants who achieved complete response (CR) and partial response (PR) based on RECIST 1.1 criteria. Complete Response (CR) for target lesion: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm. Partial Response (PR) for target lesion: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute at Milford, Milford, Massachusetts
  - Dana-Farber Cancer Institute at South Shore Hospital, Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu